CLINICAL TRIAL: NCT04115007
Title: Prostate-cancer Treatment Using Stereotactic Radiotherapy for Oligometastases Ablation in Hormone-sensitive Patients - a GETUG-AFU Phase III Randomized Controlled Trial
Brief Title: Prostate-cancer Treatment Using Stereotactic Radiotherapy for Oligometastases Ablation in Hormone-sensitive Patients
Acronym: Oligo-PRESTO
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-0160/1716; 2017-A03104-49 (Registry Identifier: ANSM)
Record Dates: First submitted 2019-10-02; First posted 2019-10-03 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Oligometastatic Hormone Sensitive Prostate Cancer
MeSH Terms: interventions — Radiosurgery; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Standard of care + Stereotactic Body Radiotherapy to oligometastases
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT) + Standard of care
- Arm B (Active Comparator): Standard of care
  Interventions: Drug: Standard of care

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy (SBRT) + Standard of care — Definition of standard of care (prior to randomization):
  * Radiotherapy to the prostate in de novo metastatic patients
  * Radiotherapy to the pelvic lymph nodes in patients with positive pelvic nodes (given as full dose to the positive lymph node and prophylactic dose to the pelvic nodal basin)
  * Long term ADT +/- intermittent treatment
  * Additional therapy following tumor board meeting : new generation hormonal therapy (abiraterone, enzalutamide, apalutamide or other approved) or chemotherapy (docetaxel).
  SBRT is delivered using the following regimen: 30 Grays (10 Gy x 3 fractions) for axial and appendicular bones and lymph node metastases if present. In case the dose cannot be safely delivered while maintaining a safe dose to the organs at risk, an alternate regimen (35 Gy in 5 fractions of 7 Gy) can be used.
  Arms: Arm A
Drug: Standard of care — Definition of standard of care (prior to randomization):
  * Radiotherapy to the prostate in de novo metastatic patients
  * Radiotherapy to the pelvic lymph nodes in patients with positive pelvic nodes (given as full dose to the positive lymph node and prophylactic dose to the pelvic nodal basin)
  * Long term ADT +/- intermittent treatment
  * Additional therapy following tumor board meeting : new generation hormonal therapy (abiraterone, enzalutamide, apalutamide or other approved) or chemotherapy (docetaxel).
  Arms: Arm B

SUMMARY:
INDICATION: Oligometastatic hormone-sensitive prostate cancer patients. METHODOLOGY: Open label, double arm, randomized 1:1, multicenter phase III study.

PRIMARY OBJECTIVE: To assess the efficacy of ablative radiotherapy (SBRT applied to all oligometastases) administered to all gross tumor sites (metastases and prostate if applicable), in oligometastatic hormone-sensitive prostate cancer patients.

ELIGIBILITY:
DIAGNOSIS AND INCLUSION CRITERIA:

1. Histologically proven adenocarcinoma of the prostate (any T stage, Gleason score, or prostate specific antigen (PSA) level);
2. Defined as M1 based on the presence of at least one bone metastasis;
3. Diagnostic workup including functional imaging (F or C-Choline-PET/CT or prostate specific membrane antigen (PSMA) PET/CT or whole body MRI) - done prior to the start of hormonal therapy;
4. With up to 5 asymptomatic or paucisymptomatic metastatic sites including at least one bone +/- pulmonary lesion +/- nodal mestastases. Are counted as a "separate" metastatic site :

   * each bone lesion, whatever the location (including pelvic localization), except if two lesions show hyperfixation in the same bone and are located < 1cm from each other they can be counted as one lesion
   * each node or nodal area located outside the true pelvis with a small diameter of 1cm or greater or with univoqual abnormal function imaging (PET Scan hyperfixation or hypersignal in whole body MRI); if multiple nodes are in close vicinity (<1cm distance between them and <4cm in total distance including the nodes, amenable to one SBRT treatment) they can be counted as one lesion
   * and patients with lung metastasis can be included
5. Patients with a previous prostatectomy or radiotherapy to the prostate and/or pelvic lymph nodes are eligible provided they have no active disease within the irradiated areas, based on functional imaging findings;
6. Age ≥18 years;
7. Eastern Cooperative Oncology Group (ECOG) ≤2;
8. Suitable for long term anti androgen therapy;
9. Patient not suitable for docetaxel or abiraterone can be included;
10. Patient that have started long term hormonal therapy are eligible if hormonal therapy has been initiated less than 2 months before randomization;
11. Patients must agree to use adequate contraception methods for the duration of study treatment and for 6 months after completing treatment;
12. Patient must have received the information sheet and signed the consent form;
13. Patients must be willing and able to comply with the protocol for the duration of the study including scheduled visits, treatment plan, laboratory tests and other study procedures;
14. Patient must be affiliated to the social security system.

NON-INCLUSION CRITERIA:

1. Patient with more than 5 metastatic sites;
2. Patient with isolated Rib hyperfixation on functional imaging without a clear correlate on morphological imaging;
3. Patient with metastatic sites other than bone, lymph nodes or lung;
4. Metastases not amenable to radiotherapy treatment with high/curative doses by multidisciplinary meeting [i.e. SBRT as per protocol or curative doses using moderate hypofractionation (55-60Gy/20) or conventional fractionation (≥74 Gy)] (e.g. gross epidural involvement, involvement of three contiguous vertebral bodies, major soft tissue involvement, and previous radiation treatment);
5. Metastases requiring immediate treatment due to significant pain (use of opioid medication), or at risk of fracture or neurological deficit;
6. Prior radiotherapy or focal ablative treatment (cryotherapy, radiofrequency ablation,…) to metastatic lesions;
7. Patients previously treated by Hormonotherapy with castrate testosterone level <50 ng/dL or ≤0.50 ng/mL or 1.73 nmol/L prior use of ADT;
8. Prior invasive (except non-melanoma skin cancer) malignancy unless disease-free for ≥5 years;
9. Contra-indication to MRI (needed for spinal SBRT);
10. Persons deprived of their liberty or under protective custody or guardianship;
11. Patients unwilling or unable to comply with the medical follow-up required by the trial because of geographic, familial, social, or psychological reasons;
12. Participation in another therapeutic trial within 30 days prior to randomization.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2020-06-23 (Actual); Primary Completion 2026-06-23 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
Castration-resistant prostate cancer free survival | From randomization to castration resistance or death from any cause, up to 1 year
  Castration-resistant prostate cancer free survival, defined as the time from randomization to castration resistance or death from any cause. Castration resistance is defined as either biochemical progression or radiological progression, with serum testosterone being at a castrated level (<50 ng/dL or <1.7 nmol/L).

SECONDARY OUTCOMES:
Overall survival | From randomization to death from any cause, up to 5 years
  The overall survival is the length of time from randomization that patients enrolled in the study are still alive. The outcome is to evaluate whether SRBT improves overall survival compared to standard of care
Prostate cancer specific survival | From randomization to death from prostate cancer, up to 5 years
  To evaluate, compared to standard of care, whether SRBT improves survival of patients until death from prostate cancer
Time to castration resistance | Time from randomization to castration resistance, up to 5 years
  The length of time patients leave without resistance to castration treatment, where deaths occurring with no castration resistance (i.e. unrelated to prostate cancer) are censored
Time to next symptomatic skeletal event | Time from randomization to the first symptomatic skeletal event, up to 5 years
  The length of time until manifestation of the first symptomatic skeletal event among the following: symptomatic bone fracture, surgery to bone or use of palliative radiotherapy to bone
Time to next symptomatic skeletal event at the treated metastatic bone sites | Time from randomization to the first symptomatic skeletal event, 5 years
  The length of time until manifestation of the first symptomatic skeletal event, at a site irradiated during the study for patients in the experimental arm, among the following: symptomatic bone fracture, the use of bone surgery, or palliative bone radiotherapy and spinal cord compression
Time to use of intermittent hormonal therapy | Time from randomization to the use of intermittent androgen deprivation therapy, up to 5 years
  The length of time patients receive continuous androgen deprivation therapy before the switch to the intermittent androgen deprivation therapy
Duration of intermittent hormonal therapy | From the end of continuous therapy to the end of intermittent therapy, up to 5 years
  The length of time patients receive intermittent androgen deprivation therapy
Time to secondary treatments (local or systemic) | From randomization to initiation of secondary treatment, up to 5 years
  The interval between the randomization and the initiation of the first treatment after disease progression: systemic chemotherapy, second line hormonal therapy, bone directed treatment (bisphosphonate or denosumab), or the use an antalgic palliative bone treatment (interventional radiology or radiotherapy)
Acute and late toxicity of stereotactic radiotherapy of oligometastases: Adverse events | Throughout study completion, up to 5 years
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale will assess the severity of sensory neuropathic disorders, this derivative into 5 grades determined by the investigator.
Severity of pain during treatment | At baseline before radiotherapy, week 6, and at every follow-up (every three months for the first three years then every 6 months for the last two years after randomization), up to 5 years
  The Brief Pain Inventory (BPI) questionnaire rapidly assesses the severity of pain and its impact on functioning. This self-report questionnaire includes:
  * A body schema
  * The maximum pain, lowest pain, usual pain within the last 15 days (Numerical Numeric rating scales (NRS) 0 to 10
  * Description of current analgesic treatment
  * An assessment of relief by a percentage scale (0-100%), Assessment of the impact of pain on: mood, relationships with others, walking, sleep, work, happiness the joy - of living, recreation, activities in general (digital scales, rating from 0 [normal] to 10 [no activity]).
The 3-level version of EQ-5D (EQ-5D-3L) questionnaire | At baseline, week 6, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, and at castration resistance (up to 5 years)
  This self-reported questionnaire that assesses the health-related quality of life of cancer patients in clinical trials consists of a descriptive system and a visual analogue scale (VAS).
  The EQ-5D-3L descriptive system comprises five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each dimension has 3 levels (1 = "no problems", 2 = "some problems", and 3 = "extreme problems"). This questionnaire provide a 5-digit score which generate a health state profile. The VAS records the patient's self-rated health on a vertical visual analogue scale where the score range from 0 (Best imaginable health state) to 100 (Worst imaginable health state). The VAS is used as a quantitative measure of health outcome that reflects the patient's own judgement.
Expanded Prostate Cancer Index Composite (EPIC) short form | At baseline, week 6, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, and at castration resistance (up to 5 years)
  This self-reported questionnaire, designed to evaluate patient function and bother after prostate cancer treatment, contains 26 item divided in 5 domains (Urinary Incontinence, Urinary Irritative/Obstructive, Bowel, Sexual, and Hormonal). Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better health-related quality of life.
Cost-effectiveness analysis of the proposed therapeutic strategy | At baseline, week 6, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, castration resistance (up to 5 years)
  To evaluate the economic cost of the SBRT treatment as compared to the treatment without radiotherapy in terms of cost assessments, incremental cost-effectiveness ratio and quality of life adjusted life years

CONTACTS AND LOCATIONS:
Overall Officials: Pierre BLANCHARD, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (35):
- France (34):
  - Institut Sainte Catherine, Avignon
  - Institut Bergonié, Bordeaux
  - Centre d'oncologie - Clinique Pasteur, Brest
  - CHRU de Brest, Brest
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Amethyst de Creil, Creil
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Institut de cancérologie de Seine et Marne - Clinique de Jossiny, Jossigny
  - Centre Oscar Lambret, Lille
  - Groupe Hospitalier Bretagne Sud, Lorient
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Azureen de Cancerologie, Mougins
  - Hôpital Privé du Confluent, Nantes
  - ICO René Gauducheau, Nantes
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - CHU Lyon Sud, Pierre-Bénite
  - CH Annecy, Pringy
  - Institut du Cancer Courlancy, Reims
  - Centre Eugene Marquis, Rennes
  - CHU de Rouen - Charles Nicole, Rouen
  - Centre Henri Becquerel, Rouen
  - Institut de cancérologie et d'hématologie universitaire de Saint Etienne, Saint-Etienne
  - CHP Saint Grégoire, Saint-Grégoire
  - HIA Begin, Saint-Mandé
  - Institut de Cancerologie Paris Nord, Sarcelles
  - Institut de cancérologie Strasbourg Europe (ICANS ), Strasbourg
  - IUCT- Oncopole -Institut Claudius Regaud, Toulouse
  - Clinique PASTEUR, Toulouse
  - Centre de radiothérapie Marie Curie de Valence, Valence
  - Centre Amethyst - Oncologie 78, Versailles
  - Gustave Roussy Cancer Campus Grand Paris, Villejuif
- CHU Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.

REFERENCES:
- [Derived] Petrelli F, Ghidini A, Ghidini M, Bukovec R, Trevisan F, Turati L, Indini A, Seghezzi S, Lonati V, Moleri G, Tomasello G, Zaniboni A. Better survival of patients with oligo- compared with polymetastatic cancers: a systematic review and meta-analysis of 173 studies. F1000Res. 2021 May 27;10:423. doi: 10.12688/f1000research.52546.4. eCollection 2021. PMID 35602670